CLINICAL TRIAL: NCT05658302
Title: Circuit-Based Deep Brain Stimulation for Parkinson's Disease P1A2&3 Catalyst
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00015253
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's disease: * Diagnosis of idiopathic PD
  * Surgery at UMN to implant DBS system with directional lead(s) and multiple independent current control IPG is planned as part of routine clinical care
  * At least 21 years old
  * Existing or planned 7T brain imagery

SUMMARY:
This study will help us better understand how the brain works in people with Parkinson's disease (PD). PD is a brain disease that gets worse over time, and affects over 10 million people world-wide. A common treatment for PD is Deep Brain Stimulation (DBS). To improve DBS therapy for PD, we need a deeper understanding of how the different parts of the brain work together in PD, and how this relates to movement and thinking problems that people with PD experience.

We may be able to use the results of this study to improve DBS treatments in the future.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurodegenerative disease affecting over 10 million people world-wide. It can be a debilitating disorder and although studied for decades, the physiological changes in the basal ganglia thalamocortical (BGTC) circuit that underlie its development remain under debate. Deep brain stimulation (DBS) of the subthalamic nucleus (STN) and internal globus pallidus (GPi) has been a highly effective therapy for many patients with PD, however, the results have been highly variable and may be associated with cognitive compromise in some patients. To advance DBS therapies for PD we require a deeper understanding of the local and network-wide circuit dynamics and their relationship to motor signs and cognitive function. This understanding will provide the rationale for optimizing STN and GPi DBS, targeting specific regions within the STN and GPi, and development of patient-specific DBS based on the patients' motor signs and cognitive profile

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD
* Surgery at UMN to implant DBS system with directional lead(s) and multiple independent current control IPG is planned as part of routine clinical care
* At least 21 years old

Exclusion Criteria:

* Other significant neurological disorder
* History of dementia
* Patients with post-operative complications or adverse effects (e.g. ON stimulation dystonias) that affect patient safety or confound the experiment will be excluded from further study
* Pregnant women
* Known radiation exposure within the last year that is determined to be unsafe when compounded with the expected radiation dose from intraoperative fluoroscopy to place ECoG strip

Min Age: 21 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: PD patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
reach-related modulation | 2 days
  reach-related modulation in beta/HFO power in DBS lead LFPs across OFF, DBS, L-dopa, and DBS+L-dopa conditions.
N-back task trials | 2 days
  directed connectivity between STN and DLPFC compared between the N-back task trials with and without stimulation.
rigidity and bradykinesia assessments | 1 day
  differences in rigidity and bradykinesia assessments between conditions: off-stimulation vs eiDBS-suppression, off-stimulation vs eiDBS-amplification, eiDBS-suppression vs eiDBS-amplification.
peak frequency of the ERs + spontaneous LFPs | 1 day
  the correlation between the peak frequency of the ERs in the GPi (or STN) and that of spontaneous LFPs in the GPi (or STN).

SECONDARY OUTCOMES:
N-back task trials | 2 days
  difference in directed connectivity between the correct reject N-back COGED trials across OFF, DBS, L-dopa, and DBS+L-dopa conditions, as well as measures of directed connectivity between STN/GPi and other ECoG sites (SC/MC/PMC/DLPFC) correlated to the N-back task trials correct response performance across the conditions mentioned above.
rigidity/bradykinesia measurements and correlations to conditions | 1 day
  correlations between each of the rigidity/bradykinesia measurements and the following: 1) amplitude of beta band oscillations in the STN or GPi and 2) information flow between the GPi (or STN) and cortical regions, and 3) PAC. Other secondary outcomes on Day 3 include 1) the coherence between ERs in the GPi or STN and ERs observed in the MC, PMC, and DLPFC; and 2) the correlation of pathway-activation measures (AFtotal) with the amplitude of ERs in the GPi (or STN) across both stimulation settings and patients.
task vs. rest and topographical location | 2 days
  task vs. rest, and topographical location, within each of the conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Minnesota, Minneapolis, Minnesota, United States